CLINICAL TRIAL: NCT02260427
Title: A Comparison of the I-gel and Self-pressurised Air-Q Intubating Laryngeal Airway (Air-Q sp) in the Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3-2014-0157
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Supraglottic Airway Device
Keywords: elective surgery; undergoing general anesthesia; elderly adult patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- the i-gel group (Experimental): After induction of general anesthesia, the i-gel will be inserted according to randomly allocated group.
  Interventions: Device: Insertion of the i-gel
- the Air-Q sp group (Active Comparator): After induction of general anesthesia, the air-Q sp will be inserted according to randomly allocated group.
  Interventions: Device: Insertion of the air-Q sp

INTERVENTIONS:
Device: Insertion of the i-gel — After induction of general anesthesia, the i-gel will be inserted according to randomly allocated group.
  Arms: the i-gel group
Device: Insertion of the air-Q sp
  Arms: the Air-Q sp group

SUMMARY:
Supraglottic airway devices (SADs) are well established in anesthetic practice. Among these devices, the i-gel has been typically widely used. The self-pressurised air-Q intubating laryngeal airway (air-Q sp) is newly developed supraglottic airway devices. It is a new single-use device that may optimise the airway sealing while reducing the potential for postoperative complications such as sore throat. The overall structure of the air-Q sp is similar to the original air-Q, except the inflatable cuff. The aim of this randomized trial was to compare the clinical performance of the i-gel and the air-Q sp in elderly patients

ELIGIBILITY:
Inclusion Criteria:

1. elderly adult patients (65-90 of age) scheduled for elective surgery undergoing general anesthesia using supraglottic airway

Exclusion Criteria:

1. Patients with a potentially difficult airway, risk of aspiration such as gastroesophageal reflux disease, or active upper respiratory tract infection

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
airway leak pressure measured after device insertion | within 5min after insertion of each device
  Airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 40 cmH2O (fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

SECONDARY OUTCOMES:
insertion parameters (insertion time and ease of insertion) | During and 1 min after insertion of each device
  Insertion time was defined as the time from the attending anesthesiologist picking up the LMA until the confirmation on capnography. Ease of insertion was graded from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Soo Kim, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research institute, Yonsei University College of Medicine, Seoul
Locations (1):
- Yonsei University College of Medicine, Gangnam Severance Hospital, 211 Eonju-ro, Gangnam-gu, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee JS, Kim DH, Choi SH, Ha SH, Kim S, Kim MS. Prospective, Randomized Comparison of the i-gel and the Self-Pressurized air-Q Intubating Laryngeal Airway in Elderly Anesthetized Patients. Anesth Analg. 2020 Feb;130(2):480-487. doi: 10.1213/ANE.0000000000003849. PMID 30320644